CLINICAL TRIAL: NCT06230094
Title: Effect of 8 Weeks Moderate & High Intensity Training on Cognitive Functions and Sleep of Female Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 014244 tabinda
Record Dates: First submitted 2023-11-24; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Sleep; Cognition

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A ( moderate intensity training) (Experimental): warm up protocol to reach maxHR 50% than moderate intensity exercise. Group A will be given moderate intensity exercise i.e brisk walk will be performed.(HR will be between 50-60%).
  Interventions: Other: moderate intensity
- Group B( high intensity training) (Experimental): warm up protocol to achieve 70% of maxHR . group Bwill be given highintensity exercise i.e skipping rope ( HR will be between 70-85%).
  Interventions: Other: high intensity

INTERVENTIONS:
Other: moderate intensity — Arm Circles, Leg Swings, Lunges, brisk walk
  Arms: Group A ( moderate intensity training)
Other: high intensity — Arm circles, Leg swings, Lunges, skipping rope
  Arms: Group B( high intensity training)

SUMMARY:
this study aims to assess ther effectiveness of moderate & high intensity training on cognitive functions and sleep of female students

DETAILED DESCRIPTION:
In group A for moderate intensity training brisk walk will be performed(HR will be between 50%- 60% of maxHR).

warmup exercise will be performed to achieve 50%HR and then brisk walk will be performed till she reaches 60%HR.

This protocol will be followed for 5days per week. In group B for high intensity training skipping rope will performed (HR will be between 70%-85% of maxHR).

warmup exercise will be performed to achieve 70%HR and then skipping rope will be performed till she reaches 85%HR.

This protocol will be followed for alternative 3days per week.

ELIGIBILITY:
Inclusion Criteria:

* female students
* age between 18- 25

Exclusion Criteria:

* History of trauma/ injury
* mental illness
* physical deformity
* infection,fever

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — age between 18-25 years
Enrollment: 32 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-03-15 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Stroop test for Cognitive Function | 8 weeks
  The Stroop Color and Word Test, interference on reading ability through three sections: word page, color page, and word-color page, each containing 5 columns with 20 items. In a 45-second timeframe, participants rapidly read words or name ink colors. Overall, the Stroop test offers a comprehensive evaluation of cognitive abilities related to interference and reading skills.
Pittsburg sleep quality index , | 8 weeks
  Each of the seven component scores, encompassing subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction, is assigned a value on a scale ranging from 0 to 3. A score of 0 signifies an absence of difficulty, while a score of 3 reflects severe difficulty within the specific component. The calculation of the Global Pittsburgh Sleep Quality Index (PSQI) score involves summing up these seven component scores, resulting in a total score that ranges from 0 to 21. Elevated global scores are indicative of lower sleep quality, and a score exceeding 5 is generally construed as suggestive of poor sleep. In terms of interpretation, a global PSQI score falling between 0 and 5 is considered representative of "good" sleep quality, while a score surpassing 5 implies a lower quality of sleep.
Digit span test | 8 weeks
  The Digit Span Test gauges short-term memory and attention span by having individuals repeat digit sequences in the same or reverse order. Scores are assigned per correctly repeated digit, with the test progressively increasing in difficulty. The total score reflects the longest accurately recalled sequences in both conditions. Interpretation reveals insights into working memory and attentional control, where a higher Digit Span Forward score signifies efficient short-term memory, while a higher Digit Span Backward score indicates superior working memory and cognitive flexibility in recalling and manipulating sequences in reverse order.
Sleep quality scale | 8 weeks
  The Sleep Quality Scale (SQS) measures sleep quality in people who live in the general population.
  Using a four-point, Likert-type scale, respondents indicate how frequently they exhibit certain sleep behaviors (0 = "few," 1 = "sometimes," 2 = "often," and 3 = "almost always"). Scores on items belong to factors 2 and 5 (restoration after sleep and satisfaction with sleep) and are reversed before being tallied. Total scores can range from 0 to 84, with higher scores demoting more acute sleep problems.

CONTACTS AND LOCATIONS:
Overall Officials: Tabinda Kanwal, Principal Investigator — Riphah International University Islamabad
Locations (1):
- Sargodha institute of health sciences, Sargodha, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No